CLINICAL TRIAL: NCT00975871
Title: Correlation of Genetic Polymorphism and Livedo Vasculitis
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Tsen-Fang Tsai/M.D, National Taiwan University Hospital
Other Study IDs: 0961172000
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2009-10-23 (Estimated); Status verified 2009-10

CONDITIONS: Livedo Vasculitis; Livedoid Vasculitis; Livedoid Vasculopathy; Genetic Pleomorphism; Leiden Mutation
Keywords: Livedo vasculitis; Genetic pleomorphism
MeSH Terms: conditions — Livedoid Vasculopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal mucosa cotton tip swab
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Livedo vasculitis is disease with recurrent courses of painful foot or ankle ulcerations, followed by healed white scars. The actual mechanism of its pathophysiology is not yet clear. It has been reported to be associated with some gene mutations, for example, factor V Leiden gene. This study is aimed to find the possible relation of these gene mutations in Taiwanese patients.

DETAILED DESCRIPTION:
Livedo vasculitis is a chronic, recurrent painful ulcerations on the ankles and feet. This chronic disease is characterized by healed white, atrophic scars named atrophie blanche. The histopathological exam on the lesion site reveals fibrin deposition within the vessel walls. It has been reported to be related to factor V Leiden mutation (heterozygous) (22.2%), prothrombin G20210A gene mutation (8.3%), PAI promotor 4G/4G genotype and methylenetetrahydrofolate reductase (MTHFR) C677T mutation in about total 30% livedo vasculitis patients. This study is trying to find the correlation between Taiwanese patients and these four genes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of livedo vasculitis

Exclusion Criteria:

* No special exclusion criteria

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsen-Fang Tsai, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan